CLINICAL TRIAL: NCT03507673
Title: Prospective, Clinical Cohort Study on the Endocrinology and Vaginal/Endometrial Microbiome of the Luteal Phase and Pregnancy After Embryo Transfer in Assisted Reproduction
Brief Title: Clinical Cohort Study on the Endocrinology and Vaginal/Endometrial Microbiome of the Luteal Phase in Assisted Reproduction
Status: Recruiting | Type: Observational
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. M.Sc. Georg Griesinger, Professor, University of Luebeck
Other Study IDs: Aktenzeichen: 18-005
Record Dates: First submitted 2018-04-14; First posted 2018-04-25 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples and Microbiological swaps (cervix uteri and endometrial sampling)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Progynova/Dydrogesterone
  Interventions: Diagnostic Test: Blood samples and microbiological swaps
- Spontaneous cycle
  Interventions: Diagnostic Test: Blood samples and microbiological swaps
- Progynova/Crinone
  Interventions: Diagnostic Test: Blood samples and microbiological swaps
- Others Medication
  Interventions: Diagnostic Test: Blood samples and microbiological swaps

INTERVENTIONS:
Diagnostic Test: Blood samples and microbiological swaps — Blood analysis and analysis of vaginal microbiota.

SUMMARY:
Rationale:

The hormone progesterone has different functions. In pregnancy, it is vital for maintenance thereof. In early pregnancy, progesterone is synthesized by the Corpus luteum (CL). Its production shifts from the CL to the placenta after several gestational weeks. This process is termed luteoplacental shift. Still, the exact time point of the luteoplacental shift remains unknown. Furthermore, the characteristics of placental progesterone increase and its relevance for the course of pregnancy has not been studied so far.

Furthermore, recent studies have shown an influence of abnormal vaginal microbiota on the likelihood to achieve and maintain pregnancy. Little is known about possible crosslinks between endocrinology and vaginal/endometrial microbiota which is why this study aims to investigate possible associations of such kind.

Objective:

The primary objective of this study is to evaluate the time point of the luteoplacental shift in patients achieving pregnancy after transfer of cryopreserved embryos subsequently to IVF/ICSI cycles. Secondary objectives are to study the characteristics of the placental progesterone increase and its function as a predictor of the course and development of pregnancies and to study vaginal/endometrial microbiota at baseline and changes associated with shift into luteal phase and early pregnancy and how this potentially relates to pregnancy outcome.

Study Design:

Prospective, multi-center, observational clinical cohort study. For the primary objective, data from a single center will be also be retrospectively analyzed.

Study population:

Female patients aged 18 to 45 years undergoing transfer of embryos after freezing and thawing 2PN oocytes or embryos.

Interventions: Blood withdrawal, vaginal/endometrial swabs and endocrine and microbiom analyses.

Study parameters/endpoints:

The main parameter is time point of progesterone increase in pregnancy in relation to initial progesterone levels by pregnancy status. Secondary, slope and magnitude of placental progesterone increase and its relevance as a predictor for the course and development of pregnancies/babies. Furthermore, vaginal microbiota of women undergoing embryo transfer and of women in early pregnancy are parameter of this study.

DETAILED DESCRIPTION:
Introduction and rationale Progesterone is a steroid hormone with different functions. In the luteal phase of the menstrual cycle elevated progesterone levels maintain the endometrium. Amongst others it stimulates glandular secretion and adjusts pattern of secreted proteins of the endometrium to provide a supportive environment for of embryo implantation. A sudden decline in progesterone levels leads to endometrial shedding and thereby menstrual bleeding. Thus, elevated progesterone levels are vital to maintain a pregnancy after successful embryo implantation. Progesterone is produced by the Corpus luteum (CL), a relict of the Graaf follicle, after ovulation in the luteal phase of the menstrual cycle and in the first weeks of pregnancy. The lifespan of the CL is assumed to be several weeks.

Before luteolysis of the CL, the production of progesterone shifts from the CL to the placenta which ensures maintenance of the pregnancy. This process is termed luteoplacental shift. Adequate placental progesterone increase is vital for the maintenance of the pregnancy and low progesterone levels can indicate inadequate development of early pregnancies. However, laboratory measurement of progesterone by conventional ELISA techniques cannot distinguish between placental progesterone and progesterone produced by the CL.

This is one reason why still little is known about the exact time point of the luteoplacental shift. In 1972 a decline of progesterone and subsequent loss of pregnancy for n=12 patients after ovariectomy or luteectomy in the 8th week of gestation but not for operations taking place in the 9th week of gestation (n= 5 patients) was reported. This is in line with in-vitro measurements from 1985 in a placental organ culture which shows the capability for progesterone production between 6th and 8th week of gestation. In 1990 it was observed in women (n=17) with absent of ovaries and constant exogenous progesterone administration achieving pregnancy by an egg donation program a significant progesterone increase in the 9th gestational week. This is in contrast to a study in a similar setting from 1991 in n=9 women who reported onset of endogenous progesterone production around the 5th week of gestation. Additionally, even the existence of the luteoplacental shift itself was questioned because of a wide range of progesterone levels observed in women achieving successful pregnancies by assisted reproduction technique (ART).

Moreover, 17-OH progesterone (17-OHP) was suspected to be produced solely by the CL in early pregnancy. This is supported by a study who found 17-OHP blood levels and vascularity of the CL decreasing from 5th till 11th week of gestation suggesting the luteoplacental shift to take place.

In summary, little is known about the exact time point of the luteoplacental shift.

Secondly, to date the slope and magnitude of the placental progesterone increase and its relevance as indicator for the latter course of the pregnancy has not been properly studied.

In routine care patients undergoing transfer of cryopreserved embryos subsequently to an IVF/ICSI cycle use estradiol and progesterone supplementation to ensure anovulation during the menstrual cycle for optimal timing of embryo transfer. For long the vaginal application of micronized progesterone have been standard of care for this purpose. In March 2017 the LOTUS I trial showed non-inferiority for oral intake (3 x 10 mg) of dydrogesterone, a retroprogesterone, a same safety profile and a higher live birth rate of approximately +5% versus micronized vaginal progesterone for patients undergoing ART. These findings are supported by a Cochrane review comprising 94 randomized trials. Therefore, in routine care the standard regime for luteal support (LPS) for all ART patients was changed to oral intake of 30 mg dydrogesterone daily at the Department of Gynecological Endocrinology and Reproductive Medicine of the University of Luebeck.

Unlike micronized progesterone the chemical properties of dydrogesterone preclude detection in laboratory progesterone measurement apart from a small fraction of cross-reactivities. This circumstance allows an analysis of endogenous progesterone despite supplementation of dihydrogesteron at the same time.

In patients undergoing transfer of cryopreserved embryos utilization of a dydrogesterone regime for LPS provides the unique opportunity to study in detail the time point and magnitude of endogenous progesterone production (i.e. the luteal shift). The choice of protocol (supplementation with exogenous sex steroids or natural cycle) is taken, when the treatment is planned based on regularity of the cycle and patient preferences.

Recent studies have shown an influence of abnormal vaginal microbiota for the prediction of pregnancy and for preclinical pregnancy loss in IVF treatment. Therefore, this study aims to investigates possible crosslinks between endocrine profile, vaginal and endometrial microbiota and the establishment and maintenance of pregnancy.

Furthermore, possible differences in vaginal bleeding pattern between different groups of cryopreservation regimes have not been evaluated so far. This study aims to investigate whether vaginal bleeding patterns might be influenced the cryopreservation regime.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 45 years
2. Transfer of cryopreserved embryos

Exclusion Criteria:

1. Fresh IVF/ICSI embryo transfer cycle
2. Evidence for ovulation on ultrasound previous to embryo transfer confirmed by a follicle ≥14mm or by a progesterone ≥1.0 µg/l in programmed cycles
3. Uterus malformations, endometrial abnormalities (on ultrasound or diagnosed by previous hysteroscopy)

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Patients attending infertility clinic.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-05-02 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Serum progesterone (microgram/Liter) levels. | 31.12. 2020

SECONDARY OUTCOMES:
Change of vaginal microbiome between follicular phase, luteal phase and early pregnancy | 31.12.2022
Vaginal bleeding pattern in the luteal phase and early pregnancy in frozen-thawed embryo transfer cycles | 31.12.2022
Association of endocrine values and bleeding, microbiome status and treatment outcome | 31.12.2022

CONTACTS AND LOCATIONS:
Overall Officials: Georg Griesinger, MD, Principal Investigator — Sektion für gynäkologische Endokrinologie und Reproduktionsmedizin
Locations (5):
- Germany (5):
  - IVF-SAAR, Saarbrücken, Saarland
  - Universitäres Kinderwunschzentrum Lübeck, Lübeck, Schleswig-Holstein
  - Universitätsklinikum Düsseldorf,UniKiD, Düsseldorf
  - Universitäres Kinderwunschzentrum, Kiel
  - University of Luebeck, Lübeck

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rommler A, Kreuzer E. [Endocrinologic aspects of habitual abortion]. Zentralbl Gynakol. 2001 Jun;123(6):344-52. doi: 10.1055/s-2001-16284. German. PMID 11488162
- [Background] Csapo AI, Pulkkinen MO, Ruttner B, Sauvage JP, Wiest WG. The significance of the human corpus luteum in pregnancy maintenance. I. Preliminary studies. Am J Obstet Gynecol. 1972 Apr 15;112(8):1061-7. doi: 10.1016/0002-9378(72)90181-0. PMID 5017636
- [Background] Ogino M. Productivity of estrogens by human placental organ culture at different stages of gestation. Endocrinol Jpn. 1985 Oct;32(5):607-13. doi: 10.1507/endocrj1954.32.607. PMID 4092668
- [Background] Devroey P, Camus M, Palermo G, Smitz J, Van Waesberghe L, Wisanto A, Wijbo I, Van Steirteghem AC. Placental production of estradiol and progesterone after oocyte donation in patients with primary ovarian failure. Am J Obstet Gynecol. 1990 Jan;162(1):66-70. doi: 10.1016/0002-9378(90)90822-o. PMID 2154102
- [Background] Scott R, Navot D, Liu HC, Rosenwaks Z. A human in vivo model for the luteoplacental shift. Fertil Steril. 1991 Sep;56(3):481-4. doi: 10.1016/s0015-0282(16)54544-0. PMID 1894025
- [Background] Azuma K, Calderon I, Besanko M, MacLachlan V, Healy DL. Is the luteo-placental shift a myth? Analysis of low progesterone levels in successful art pregnancies. J Clin Endocrinol Metab. 1993 Jul;77(1):195-8. doi: 10.1210/jcem.77.1.7686913.
- [Background] Tulchinsky D, Simmer HH. Sources of plasma 17alpha-hydroxyprogesterone in human pregnancy. J Clin Endocrinol Metab. 1972 Dec;35(6):799-808. doi: 10.1210/jcem-35-6-799. No abstract available. PMID 4634481
- [Background] Jarvela IY, Ruokonen A, Tekay A. Effect of rising hCG levels on the human corpus luteum during early pregnancy. Hum Reprod. 2008 Dec;23(12):2775-81. doi: 10.1093/humrep/den299. Epub 2008 Aug 10. PMID 18694877
- [Background] Tournaye H, Sukhikh GT, Kahler E, Griesinger G. A Phase III randomized controlled trial comparing the efficacy, safety and tolerability of oral dydrogesterone versus micronized vaginal progesterone for luteal support in in vitro fertilization. Hum Reprod. 2017 May 1;32(5):1019-1027. doi: 10.1093/humrep/dex023. PMID 28333318
- [Background] van der Linden M, Buckingham K, Farquhar C, Kremer JA, Metwally M. Luteal phase support for assisted reproduction cycles. Cochrane Database Syst Rev. 2015 Jul 7;2015(7):CD009154. doi: 10.1002/14651858.CD009154.pub3. PMID 26148507
- [Background] Haahr T, Jensen JS, Thomsen L, Duus L, Rygaard K, Humaidan P. Abnormal vaginal microbiota may be associated with poor reproductive outcomes: a prospective study in IVF patients. Hum Reprod. 2016 Apr;31(4):795-803. doi: 10.1093/humrep/dew026. Epub 2016 Feb 23. PMID 26911864
- [Background] van Oostrum N, De Sutter P, Meys J, Verstraelen H. Risks associated with bacterial vaginosis in infertility patients: a systematic review and meta-analysis. Hum Reprod. 2013 Jul;28(7):1809-15. doi: 10.1093/humrep/det096. Epub 2013 Mar 29. PMID 23543384
- [Background] Graspeuntner S, Bohlmann MK, Gillmann K, Speer R, Kuenzel S, Mark H, Hoellen F, Lettau R, Griesinger G, Konig IR, Baines JF, Rupp J. Microbiota-based analysis reveals specific bacterial traits and a novel strategy for the diagnosis of infectious infertility. PLoS One. 2018 Jan 9;13(1):e0191047. doi: 10.1371/journal.pone.0191047. eCollection 2018. PMID 29315330
- [Result] Gellersen B, Brosens JJ. Cyclic decidualization of the human endometrium in reproductive health and failure. Endocr Rev. 2014 Dec;35(6):851-905. doi: 10.1210/er.2014-1045. Epub 2014 Aug 20. PMID 25141152
- [Result] Di Renzo GC, Giardina I, Clerici G, Brillo E, Gerli S. Progesterone in normal and pathological pregnancy. Horm Mol Biol Clin Investig. 2016 Jul 1;27(1):35-48. doi: 10.1515/hmbci-2016-0038. PMID 27662646
- [Derived] Eggersmann TK, Hamala N, Hiller AR, Depenbusch M, Schultze-Mosgau A, Edimiris P, Baston-Bust D, Bielfeld AP, Kruessel JS, von Otte S, Junkers W, Tauchert S, Vonthein R, Griesinger G. Live birth rates are unrelated to sex-steroid levels on ET day in a dydrogesterone-based 'programmed-ovulatory FET' protocol: a multi-centric prospective cohort study. Hum Reprod Open. 2025 Sep 15;2025(4):hoaf058. doi: 10.1093/hropen/hoaf058. eCollection 2025. PMID 41221299
- [Derived] Neumann K, Masuch A, Vonthein R, Depenbusch M, Schultze-Mosgau A, Eggersmann TK, Griesinger G. Dydrogesterone and 20alpha-dihydrodydrogesterone plasma levels on day of embryo transfer and clinical outcome in an anovulatory programmed frozen-thawed embryo transfer cycle: a prospective cohort study. Hum Reprod. 2022 May 30;37(6):1183-1193. doi: 10.1093/humrep/deac045. PMID 35323905